CLINICAL TRIAL: NCT00481572
Title: Continuous Terlipressin Versus Vasopressin Infusion in Septic Shock. A Randomized, Controlled, Pilot Trial. "THE TERLIVAP STUDY"
Brief Title: Continuous Infusion of Terlipressin in Septic Shock
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Andrea Morelli, University of Roma "La Sapienza"
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1124
Record Dates: First submitted 2007-05-30; First posted 2007-06-01 (Estimated); Last update posted 2008-02-29 (Estimated); Status verified 2008-02

CONDITIONS: Septic Shock
Keywords: Sepsis; Septic Shock; vasopressin; terlipressin
MeSH Terms: conditions — Shock, Septic; Sepsis; Diabetes Insipidus | interventions — Terlipressin; Vasopressins; Norepinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Terlipressin
  Interventions: Drug: Terlipressin
- 2 (Experimental): Vasopressin
  Interventions: Drug: Vasopressin
- 3 (Active Comparator): titrated norepinephrine
  Interventions: Drug: Norepinephrine

INTERVENTIONS:
Drug: Terlipressin — continuous terlipressin infusion 1.3 µg•kg-1 over a period of 48 hrs
  Arms: 1
Drug: Vasopressin — continuous intravenous infusion of vasopressin 0.03 U•min-1 over a period of 48 hrs
  Arms: 2
Drug: Norepinephrine — titrated norepinephrine over a period of 48 hrs
  Arms: 3

SUMMARY:
The purpose of this study is to determine whether: A)the continuous infusion ultra-low dose of terlipressin (1.3 micrograms/kg/h) is able to stabilize hemodynamic in patients with septic shock, reducing the risk of adverse effects related to the bolus dose.B)the continuous infusion ultra-low dose of terlipressin may be use in lieu of vasopressin.

DETAILED DESCRIPTION:
Forty-five septic shock patients requiring vasopressor support to maintain mean arterial pressure between 65 and 75 mmHg despite adequate volume resuscitation were enrolled in the study. Patients were randomly allocated to be treated with either a) a continuous terlipressin infusion (1.3 µg•kg-1), b) vasopressin (0.03 U•min-1), or c) titrated norepinephrine (control; each n = 15). In both the terlipressin and vasopressin group, norepinephrine was additionally administered to achieve a mean arterial pressure (MAP) between 65 and 75 mmHg, if necessary. Data from right heart catheterization, thermo-dye dilution catheter, gastric tonometry as well as data from organ function, cytokines concentrations, were obtained at baseline and after 12, 24, 36 and 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Septic shock
* vasopressor support to maintain mean arterial pressure (MAP) between 65 and 75 mmHg despite adequate volume resuscitation (pulmonary artery occlusion pressure = 13-18 mmHg and central venous pressure = 8-12 mmHg)

Exclusion Criteria:

* Pregnancy
* Present cardiac dysfunction
* Present or suspected acute mesenteric ischemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2007-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Systemic and regional hemodynamics | during the first 48 hours from the onset of septic shock

SECONDARY OUTCOMES:
Markers of inflammation,organ functions,adverse effects. | during the first 48 hours from the onset of septic shock

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Morelli, MD, Study Director — Departement of Anesthesiology and Intensive Care of the University of Rome "La Sapienza"
Locations (1):
- Department of Anesthesiology and Intensive care of the University of Rome "La Sapienza", Rome, Viale Del Policlinico 155, Italy

REFERENCES:
- [Derived] Morelli A, Ertmer C, Rehberg S, Lange M, Orecchioni A, Cecchini V, Bachetoni A, D'Alessandro M, Van Aken H, Pietropaoli P, Westphal M. Continuous terlipressin versus vasopressin infusion in septic shock (TERLIVAP): a randomized, controlled pilot study. Crit Care. 2009;13(4):R130. doi: 10.1186/cc7990. Epub 2009 Aug 10. PMID 19664253